CLINICAL TRIAL: NCT04772534
Title: A Phase 3, Open-label Clinical Study to Evaluate the Immunogenicity and Safety of 9vHPV Vaccine, in Japanese Boys and Girls, 9 to 15 Years of Age.
Brief Title: Immunogenicity and Safety of the 9-valent Human Papillomavirus (9vHPV) Vaccine in Japanese Boys and Girls (V503-066)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-066; V503-066 (Other: MSD); jRCT2031210080 (Registry Identifier: jRCT); 2020-001170-29 (EudraCT Number)
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 3-dose in 9 to 15 year old boys (Experimental): 9 to 15 year old boys will receive a 3-dose regimen of 9vHPV vaccine (Day 1, Month 2 and Month 6).
  Interventions: Biological: 9vHPV vaccine
- 2-dose in 9 to 14 year old boys (Experimental): 9 to 14 year old boys receive a 2-dose regimen of 9vHPV vaccine (Day 1 and Month 6).
  Interventions: Biological: 9vHPV vaccine
- 2-dose in 9 to 14 year old girls (Experimental): 9 to 14 year old girls receive a 2-dose regimen of 9vHPV vaccine (Day 1 and Month 6).
  Interventions: Biological: 9vHPV vaccine

INTERVENTIONS:
Biological: 9vHPV vaccine — 9-valent human papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) administered as a 0.5-mL intramuscular injection
  Other Names: V503; SILGARD®9; GARDASIL™9

SUMMARY:
The primary objective of this study is the estimation of the human papillomavirus (HPV) 6, 11, 16, 18, 31, 33, 45, 52 and 58 seroconversion at 1 month post last dose (Month 7) following 3 doses and 2 doses of the 9-valent human papillomavirus (9vHPV) vaccine. No hypothesis will be tested since this study is an estimation-only study.

ELIGIBILITY:
Inclusion Criteria:

* Is Japanese male or female.
* Is aged at the time of providing the documented informed consent (inclusive): (3-dose boy arm) male from 9 years to 15 years old, (2-dose boy arm) male from 9 years to 14 years old, or (2-dose girl arm) female from 9 years to 14 years old.
* Has a legally acceptable representative who can read, understand and complete the vaccination report card (VRC).
* Has not yet had coitarche and does not plan on becoming sexually active during the Day 1 through Month 7.

Exclusion Criteria:

* Has a fever (defined as oral temperature ≥37.5°C) within the 24-hour period prior to the Day 1 visit.
* Has a history of severe allergic reaction that required medical intervention.
* Is allergic to any vaccine component, including aluminum, yeast, or Benzonase™.
* Has known thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Is currently immunocompromised or has been diagnosed as having a congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other auto immune condition.
* Has a history of splenectomy.
* Has a history of genital warts or positive test for human papillomavirus (HPV).
* Is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within 12 months) of drug or alcohol abuse or dependence at the discretion of the investigator. .
* Has received within 12 months prior to enrollment, is receiving, or plans to receive during Day 1 through Month 7 of the study, any study-prohibited concomitant immunosuppressive therapy .
* Has received within the 3 months prior to the Day 1 vaccination, is receiving, or plans to receive during Day 1 through Month 7 of the study, any immune globulin product or blood-derived product other than intravenous gamma globulin (IVIG).
* Has received inactivated or recombinant vaccines within 14 days prior to Day 1 vaccination or receipt of live vaccines within 28 days prior to Day 1 vaccination.
* Has previously received a marketed HPV vaccine or has participated in a clinical trial for any HPV vaccine (receiving either active agent or placebo).
* Is concurrently enrolled in other clinical studies of investigational agents.
* Is unlikely to adhere to the study procedures, keep appointments, or is planning to permanently relocate from the area prior to the completion of the study or to leave for an extended period when study visits would need to be scheduled.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (12):
- Japan (12):
  - Sotobo Children's Clinic ( Site 6616), Isumi, Chiba
  - Ohigesenseino Kodomo Clinic ( Site 6607), Sapporo, Hokkaido
  - Motomachi Pediatric Clinic ( Site 6606), Sapporo, Hokkaido
  - Medical Corporation Bunmeikai Okuda E.N.T ( Site 6611), Sakai, Osaka
  - Fukui General Hospital ( Site 6614), Fukui
  - Nomura Clinic Namba ( Site 6608), Osaka
  - Medical Corporation Kanyukai Kikumori Otolaryngology Clinic ( Site 6612), Osaka
  - Doujin Memorial Medical Foundation, Meiwa Hospital ( Site 6603), Tokyo
  - Okawa Children & Family Clinic ( Site 6610), Tokyo
  - Shinjuku Higashiguchi Clinic ( Site 6602), Tokyo
  - Hayashi Clinic ( Site 6615), Tokyo
  - Ogikuboekimae Clinic ( Site 6601), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 12 centers in Japan.
Groups:
- 3-Dose Regimen: 9 to 15 Year Old Boys: 9 to 15 year old boys received a 3-dose regimen of 9-valent human papillomavirus (9vHPV) vaccine (Day 1, Month 2 and Month 6).
- 2-dose Regimen: 9 to 14 Year Old Boys: 9 to 14 year old boys received a 2-dose regimen of 9vHPV vaccine (Day 1 and Month 6).
- 2-dose Regimen: 9 to 14 Year Old Girls: 9 to 14 year old girls received a 2-dose regimen of 9vHPV vaccine (Day 1 and Month 6).
Period: Overall Study
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Girls
Started | 105 | 104 | 105
Completed | 101 | 104 | 104
Not Completed | 4 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 3-Dose Regimen: 9 to 15 Year Old Boys: 9 to 15 year old boys received a 3-dose regimen of 9vHPV vaccine (Day 1, Month 2 and Month 6).
- Total: Total of all reporting groups
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Girls | Total
Number analyzed (Participants) | 105 | 104 | 105 | 314
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.8 (2.0) | 11.5 (1.7) | 11.4 (1.6) | 11.6 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 105 | 105
  Male | 105 | 104 | 0 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 105 | 104 | 105 | 314
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 105 | 104 | 105 | 314
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Percentages for the HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58
Description: The percentage of seropositive participants is reported. Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined using competitive Luminex Immunoassay (cLIA). Seroconversion was defined as changing serostatus from seronegative at Day 1 to seropositive at 4 weeks post last vaccination.
Time Frame: 1 month after final dose (Month 7)
Population: All participants who received all 9vHPV vaccinations at the correct dose and day range, have provided blood samples for serology within 21 to 49 days of the last dose, are seronegative to the appropriate HPV type(s) at Day 1, and had no protocol violations that could interfere with immune response, are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Girls
Number analyzed (Participants) | 103 | 104 | 104
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 90 | 91 | 93
  Anti-HPV 6 | 100.0 [96.0 to 100.0] | 100.0 [96.0 to 100.0] | 100.0 [96.1 to 100.0]
  Anti-HPV 11: number analyzed (Participants) | 90 | 91 | 93
  Anti-HPV 11 | 100.0 [96.0 to 100.0] | 100.0 [96.0 to 100.0] | 100.0 [96.1 to 100.0]
  Anti-HPV 16: number analyzed (Participants) | 98 | 98 | 97
  Anti-HPV 16 | 100.0 [96.3 to 100.0] | 100.0 [96.3 to 100.0] | 100.0 [96.3 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 94 | 92 | 83
  Anti-HPV 18 | 100.0 [96.2 to 100.0] | 100.0 [96.1 to 100.0] | 100.0 [95.7 to 100.0]
  Anti-HPV 31: number analyzed (Participants) | 90 | 93 | 90
  Anti-HPV 31 | 100.0 [96.0 to 100.0] | 100.0 [96.1 to 100.0] | 100.0 [96.0 to 100.0]
  Anti-HPV 33: number analyzed (Participants) | 85 | 90 | 96
  Anti-HPV 33 | 100.0 [95.8 to 100.0] | 100.0 [96.0 to 100.0] | 100.0 [96.2 to 100.0]
  Anti-HPV 45: number analyzed (Participants) | 94 | 95 | 99
  Anti-HPV 45 | 100.0 [96.2 to 100.0] | 100.0 [96.2 to 100.0] | 100.0 [96.3 to 100.0]
  Anti-HPV 52: number analyzed (Participants) | 97 | 96 | 97
  Anti-HPV 52 | 100.0 [96.3 to 100.0] | 100.0 [96.2 to 100.0] | 100.0 [96.3 to 100.0]
  Anti-HPV 58: number analyzed (Participants) | 101 | 100 | 99
  Anti-HPV 58 | 100.0 [96.4 to 100.0] | 100.0 [96.4 to 100.0] | 100.0 [96.3 to 100.0]

2. Primary Outcome: Number of Participants With at Least 1 Injection-site Adverse Event (AE)
Description: The number of participants with injection-site AEs (erythema/redness, pain and swelling) is reported. An AE any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to 5 days after each vaccination (up to ~6 months)
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Groups:
- 2-dose in 9 to 14 Year Old Boys: 9 to 14 year old boys received a 2-dose regimen of 9vHPV vaccine (Day 1 and Month 6).
- 2-dose in 9 to 14 Year Old Girls: 9 to 14 year old girls received a 2-dose regimen of 9vHPV vaccine (Day 1 and Month 6).
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose in 9 to 14 Year Old Boys | 2-dose in 9 to 14 Year Old Girls
Number analyzed (Participants) | 103 | 104 | 104
Participants | 87 | 85 | 92

3. Primary Outcome: Number of Participants With at Least 1 Systemic Adverse Event
Description: The number of participants with a systemic AE is reported. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to 15 days after each vaccination (up to ~6.5 months)
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose in 9 to 14 Year Old Boys | 2-dose in 9 to 14 Year Old Girls
Number analyzed (Participants) | 103 | 104 | 104
Participants | 55 | 41 | 33

4. Primary Outcome: Number of Participants With at Least 1 Serious Adverse Event (SAE)
Description: The number of participants with an SAE is reported. An SAE is defined as one that results in death, is life threatening, or requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or other important medical event that may require medical intervention.
Time Frame: Up to ~Month 30
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Girls
Number analyzed (Participants) | 103 | 104 | 104
Participants | 0 | 2 | 3

5. Secondary Outcome: Geometric Mean Titers (GMTs) for the HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58
Description: The GMT for each HPV serotype is presented. Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined using competitive Luminex Immunoassay (cLIA).
Time Frame: 1 month after final dose (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: GMT (mMU/mL)
Groups:
- 3-Dose Regimen: 9 to 15 Year Old Boys: 9 to 15 year old boys received a 3-dose regimen of 9vHPV vaccine (Day 1, Month 2 and Month 6).).
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Girls
Number analyzed (Participants) | 103 | 104 | 104
GMT (mMU/mL)
  Anti-HPV 6: number analyzed (Participants) | 90 | 91 | 93
  Anti-HPV 6 | 1759.8 [1481.2 to 2090.8] | 2417.0 [2057.3 to 2839.6] | 2343.2 [2036.1 to 2695.5]
  Anti-HPV 11: number analyzed (Participants) | 90 | 91 | 93
  Anti-HPV 11 | 1341.8 [1136.1 to 1584.9] | 1510.1 [1310.3 to 1740.4] | 1508.5 [1340.8 to 1697.0]
  Anti-HPV 16: number analyzed (Participants) | 98 | 98 | 97
  Anti-HPV 16 | 7020.8 [5955.3 to 8277.1] | 9808.5 [8437.7 to 11402.0] | 9800.0 [8440.1 to 11379.1]
  Anti-HPV 18: number analyzed (Participants) | 94 | 92 | 83
  Anti-HPV 18 | 2629.6 [2154.7 to 3209.1] | 2464.6 [2095.6 to 2898.5] | 2999.8 [2509.3 to 3586.3]
  Anti-HPV 31: number analyzed (Participants) | 90 | 93 | 90
  Anti-HPV 31 | 2095.0 [1717.2 to 2555.9] | 1908.5 [1619.3 to 2249.4] | 1838.7 [1571.8 to 2151.0]
  Anti-HPV 33: number analyzed (Participants) | 85 | 90 | 96
  Anti-HPV 33 | 894.9 [753.1 to 1063.4] | 1272.1 [1085.2 to 1491.2] | 1283.1 [1132.4 to 1453.8]
  Anti-HPV 45: number analyzed (Participants) | 94 | 95 | 99
  Anti-HPV 45 | 848.9 [701.1 to 1027.8] | 508.4 [431.7 to 598.8] | 599.6 [520.6 to 690.4]
  Anti-HPV 52: number analyzed (Participants) | 97 | 96 | 97
  Anti-HPV 52 | 925.3 [774.9 to 1105.0] | 587.4 [503.3 to 685.5] | 582.7 [517.3 to 656.4]
  Anti-HPV 58: number analyzed (Participants) | 101 | 100 | 99
  Anti-HPV 58 | 1401.7 [1177.4 to 1668.8] | 1350.6 [1155.1 to 1579.1] | 1379.8 [1216.4 to 1565.1]

ADVERSE EVENTS:
Time Frame: Up to ~Month 30
Description: All treated participants are included.
Arm/Group | 3-Dose Regimen: 9 to 15 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Boys | 2-dose Regimen: 9 to 14 Year Old Girls
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/104 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/103 | 2/104 | 3/104
Other Adverse Events (participants affected / at risk) | 18/103 | 12/104 | 8/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3-Dose Regimen: 9 to 15 Year Old Boys (N=103) | 2-dose Regimen: 9 to 14 Year Old Boys (N=104) | 2-dose Regimen: 9 to 14 Year Old Girls (N=104)
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3-Dose Regimen: 9 to 15 Year Old Boys (N=103) | 2-dose Regimen: 9 to 14 Year Old Boys (N=104) | 2-dose Regimen: 9 to 14 Year Old Girls (N=104)
Pyrexia (General disorders) | 18 | 12 | 8
Headache (Nervous system disorders) | 10 | 9 | 6
Nasopharyngitis (Infections and infestations) | 6 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT04772534/Prot_SAP_000.pdf